CLINICAL TRIAL: NCT06334718
Title: A Mixed-methods Evaluation of Integrating Drone-delivered Automated External Defibrillators Into the Ambulance Service Response to Out-of-hospital Cardiac Arrest
Brief Title: Drone Delivered Defibrillators (The 3D Project).
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Collaborators: Welsh Ambulance Service NHS Trust (Unknown)
Responsible Party: Principal Investigator, Keith Couper, Associate Professor, University of Warwick
Other Study IDs: 318417; NIHR204382 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2024-03-18; First posted 2024-03-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: Defibrillators; Unmanned Aerial Devices; Heart Arrest; Cardiac Arrest, Out-of-Hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Interviews and simulation — Work package 1: interview study Work package 2: simulated cardiac arrest study with AED delivered by drone following a simulated emergency (999) call.

SUMMARY:
The goal of this observational study is to explore the optimisation and integration of a drone-delivered Automated External Defibrillator (AED) system into the pre-hospital response to out-of-hospital cardiac arrest. The study is being conducted by the University of Warwick and Welsh Ambulance Service National Health Service Trust (both in the UK)

There are two separate packages of work. In work package 1 the investigators will interview people who have been involved in emergency (999) calls for cardiac arrest, asking them about their experiences with the call-handler and how they feel they might have responded if they had received an AED that had been delivered by a flying drone.

In work package 2 the investigators will conduct simulated cardiac arrests. The participants in the study will make an emergency (999) call to a trained call-handler and, once the cardiac arrest is identified during the call, a drone will be activated from a distant location and fly up to 2km to the test site and deliver an AED. The investigators will record how long it takes to retrieve and attach the AED, and ask the participants for their views about the interaction with the call-handler, AED and drone.

DETAILED DESCRIPTION:
Background and study aims

Only 10% people survive after having a cardiac arrest in the community. Delivering an electric shock to the heart using a defibrillator greatly improves someone's chance of surviving.

Automated External Defibrillators (AEDs) are a type of defibrillator that may be found in public places. You can attach an AED to someone who is having a cardiac arrest. The AED may give them an electric shock and help their heart beat normally again. They are safe for members of the public to use, even if they are not trained to use them.

However, if a person is helping someone who has had a cardiac arrest it may be very difficult to find a nearby AED soon enough to make a real difference. There may be better ways to deliver AEDs quickly to more people who need them. In Sweden, ambulance services use flying drones to deliver AEDs to people after cardiac arrest. Nobody has yet demonstrated how the investigators will do this in the UK.

This study aims to explore the optimisation and integration of a drone-delivered AED system into the pre-hospital response to out-of-hospital cardiac arrest, as a necessary pre-requisite to real-life flight operations.

What does the study involve?

The investigators will build a fully-functioning system to deliver an Automated External Defibrillator using a flying drone to someone who has had a cardiac arrest.

The study has two main parts:

Part one - interview study

1. The investigators will ask people who have previously used an AED in real-life cardiac arrests about their experiences. The investigators will ask them what they think about how a drone bringing them an AED might have helped them at the time.
2. The investigators will analyse their responses using the Theoretical Domains Framework, which links to the COM-B (Capability, Opportunity and Motivation - Behaviour) framework and the BCW (Behaviour Change Wheel). This will allow the investigators to identify the main barriers and facilitators to drone-delivery of AEDs, and to determine interventions to overcome them and policies to help with the implementation of these interventions.
3. This work will help determine how to optimise future real-world drone-delivered AED systems

The investigators will recruit primarily through Welsh Ambulance Service NHS Trust's existing contacts with cardiac arrest survivor and bystander groups, but will also recruit via the social media platforms of Welsh Ambulance Service NHS Trust and Warwick University. The investigators will approach national charities with whom we have existing relationships (Resuscitation Council UK, British Heart Foundation and Sudden Cardiac Arrest UK) to help with study advertisement if required.

This will be a semi-structured interview conducted remotely, either using Microsoft TEAMS or, if the participant prefers, over the phone. The investigators will interview a mix of people who did and did not use an AED during their cardiac arrest experience. Interviews will last up to 45 minutes and will be audio-recorded before being sent to a University-approved transcription company for transcription. The participant information sheet provides information about support for participants should the interview process and talking about this sensitive topic prove difficult for them. All audio files and transcripts will be stored on a University of Warwick-managed computer, in an encrypted folder.

A senior research fellow will conduct and analyse the interviews, with assistance from the Chief Investigator. The investigators will perform a framework analysis using the Theoretical Domains Framework (TDF) to identify barriers and facilitators to drone-delivered AED use and to effective interaction with the 999 call-handler.

The investigators will group the 14 domains of the TDF so that we can characterise barriers and facilitators to effective use of a drone-delivered AED according to a bystander's 'Capability', 'Opportunity' and 'Motivation' - the so-called COM-B (Capability, Opportunity, Motivation - Behaviour) framework (38). We will then map the three core targets for behavioural change to identify potential interventions to enact this change using the Behaviour Change Wheel.

The key outcomes are a list of barriers and facilitators to drone-delivered AED use, and a list of potential interventions (for future testing or implementation) to optimise the future use of drone-delivered AEDs in the real-world cardiac arrest response.

Part two - test flights and simulated cardiac arrests

1. The investigators will show that a drone can effectively and safely make a long-distance ('beyond visual-line-of-sight', or BVLOS) flight carrying an AED.
2. The investigators will integrate drone systems with ambulance systems. The investigators will show how the investigators can automatically and quickly activate a drone after an emergency (999) call is made about a cardiac arrest.
3. The investigators will develop real-time communication systems between drone pilots and the ambulance service during flight.
4. The investigators will perform test flights:

   * A participant in our research study will find a simulated cardiac arrest patient (a resuscitation manikin) and make an emergency (999) call.
   * The ambulance service will activate the drone and the investigators will test how effective the entire system works from the start of the emergency (999) call to final delivery of the AED.
   * The investigators will record key timings including flight timings, and how long it takes the participant to retrieve and then apply the AED
   * The investigators will review audio recordings of the mock emergency (999) calls and video from the drone and from the simulation site to identify additional information about how the participants interacted with the drone and with the AED.

The simulations will be performed in an outdoor location, and at a site where investigators can control access. The drone will fly 'beyond visual line of sight' up to 2km away from the cardiac arrest site. The 'patient' will be a manikin, but in all other respects the simulation will run as the investigators envisage a real-world cardiac arrest call would: the 999 call goes through to a trained operator (at a training centre), following established cardiac arrest scripts and, once cardiac arrest is diagnosed, the communication processes with the remote drone operator will occur in real-time.

Members of the study team will be on hand to make timings and to administer a post-simulation questionnaire (based on a 'System Usability Scale', to gauge how the participant found the interaction with the drone) and to conduct a brief (<5 min) interview to record their thoughts on the process, particularly the interaction with drone and call-handler.

Audio and visual recordings will be securely transferred in electronic format to the Chief Investigator, who will store them in a University of Warwick managed computer, in an encrypted folder.

Key outcomes are:

* Time from start of emergency (999) call and diagnosis of cardiac arrest to drone having started flight
* Total flight time
* Time from drone arrival at scene and when it is safe for participant to retrieve AED. (AED will be lowered by winch to the ground. The call-handler will have real-time communications with the drone operator and will be informed when it is safe to approach - they will then inform the participant)
* Total time from emergency call to AED application and (simulated) shock
* Hands off CPR time (time from stopping CPR to retrieve AED to time that CPR starts again after AED has been applied and delivered a (simulated) shock
* Time that participant spends away from the patient's side (retrieving the AED)

Where is the study run from?

The study is run by researchers at the University of Warwick, UK, in collaboration with Welsh Ambulance Service National Health Service Trust and a commercial drone company (SkyBound Rescuer, Southampton, UK). All three organisations are based in the United Kingdom

When is the study starting and how long is it expected to run for?

Development work on the system began on 1st May 2023. The investigators will recruit to the interview study in April and May 2024, and perform the cardiac arrest simulations in August 2024. The study analyses will be completed by 31st October 2024.

Who is funding the study?

The National Institute for Health and Care Research (NIHR) Research for Patient Benefit (RfPB) scheme. Health and Care Research Wales are supporting excess treatment costs. Both are organisations in the UK.

ELIGIBILITY:
Inclusion Criteria (interviews):

* have mental capacity to make decisions about study participation.
* have provided bystander interventions (CPR +/- use of an AED) during an out-of-hospital cardiac arrest
* are able to conduct interviews in English.
* are willing to have an audio recording made of the interview.

Exclusion Criteria (interviews):

* Those who have not previously provided any bystander intervention during an out-of-hospital cardiac arrest
* (in the judgement of the interviewer, are not able to understand or communicate effectively in English.)
* Those who do not agree to be audio recorded

Inclusion Criteria (simulation):

* aged 18 years of age or older
* have mental capacity to make decisions about study participation.
* believe themselves to have the physical and mental capability to perform CPR and use an AED in an outdoor environment.
* believe themselves able to use a mobile phone to communicate with a 999 call-handler.

Exclusion Criteria (simulation):

* those who are or who believe themselves to be pregnant
* those that are unable to complete the simulation because of physical or psychological distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers. For interviews the investigators will recruit from people who meet the eligibility criteria and who have previously agreed to have their contact details held by Welsh Ambulance Service. For the simulation study the investigators will recruit members of the public from local community groups near to the site of the simulation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Time away from patient's side (SIMULATION) | During simulation procedure (cardiac arrest scenario)
  Time from leaving patient to retrieve drone-delivered AED to returning to patient's side with AED
Barriers and facilitators to drone-delivered AED use (INTERVIEW) | Following analysis and synthesis of all interviews (24 planned), April 2024 to October 2024
  Findings from interview, after analysis using theoretically-informed frameworks

SECONDARY OUTCOMES:
Interventions to overcome barriers to drone delivered AED use (INTERVIEW) | Following analysis and synthesis of all interviews (24 planned); April 2024 to October 2024
  List of interventions, informed by behavioural change models and techniques, to overcome barriers identified in interviews
Hands off CPR time (SIMULATION) | During simulation procedure (cardiac arrest scenario)
  Time from stopping CPR to starting CPR again after the AED has been attached and delivered a shock
Total time from start of 999 call to AED application and first shock (SIMULATION) | During simulation procedure (cardiac arrest scenario)
  Total time from start of 999 call to AED application (and first shock), in mins:secs
Total drone flight time (SIMULATION) | During simulation procedure (cardiac arrest scenario)
  From start of flight to delivery of AED to scene
Time from drone arrival to safe to approach (SIMULATION) | During simulation procedure (cardiac arrest scenario)
  Time from drone arrival at scene and when it is safe for participant to retrieve AED. (AED will be lowered by winch to the ground. The call-handler will have real-time communications with the drone operator and will be informed when it is safe to approach - they will then inform the participant)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Smith, MBChB, PhD, Principal Investigator — University of Warwick
Locations (1):
- University of Warwick, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Interviews: Key codes and themes that emerge during interview analysis. Anonymised individualised quotes may appear in published work.
  Simulation: simulation timings, key findings from review of audio and video analyses and post-event review.
Supporting Information: Study Protocol
Time Frame: Data will be available from time of open-access peer-reviewed publication - one each planned for interview and for simulation study.
  Protocol available from time of project registration
Access Criteria: No restrictions
URL: https://www.fundingawards.nihr.ac.uk/award/NIHR204382

DOCUMENTS (1):
  • Study Protocol (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT06334718/Prot_000.pdf